CLINICAL TRIAL: NCT01117805
Title: Women of Color and Asthma Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Randall Brown, PI, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R18HL094272-01 (NIH)
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Subjects will be randomized to the program intervention which is a female-specific, culturally relevant, self-regulation based telephone counseling intervention designed for African American women with asthma.
  Interventions: Behavioral: Telephone counseling intervention
- usual care (No Intervention): Usual care at the University of Michigan Health System is based on the guidelines as recommended by the National Asthma Education and Prevention Program Expert Panel Report 3 (NAEPP-EPR3): Diagnosis and Treatment of Asthma and is coordinated so that all patients receive the same action plan, educational materials and instructions in use of devices.

INTERVENTIONS:
Behavioral: Telephone counseling intervention — self-regulation telephone counseling program for African American women with asthma
  Other Names: Women Breathe Free
  Arms: Intervention

SUMMARY:
The proposed randomized controlled trial will evaluate an innovative intervention in 420 African American women with asthma. It will be the first to use a highly tailored, telephone counseling approach to address both specific cultural factors affecting asthma and the influence of female sex and gender on control.

DETAILED DESCRIPTION:
Research and practice efforts in asthma continue to overlook one of the most vulnerable subgroups of Americans, minority women. Women of color, especially African Americans, bear a significantly disproportionate burden of asthma among adults. However, no rigorous trial of an intervention to assist them with their particular challenges can be located. The proposed randomized controlled trial will evaluate an innovative intervention in 420 African American women with asthma. It will be the first to address both specific cultural factors affecting asthma and the influence of female sex and gender on control. It will use a highly tailored, telephone counseling approach designed to foster partnership with the clinician, resolution of specific asthma management problems, and identification of important contributing influences often misunderstood or ignored by women themselves as well as the health care system. It will attend closely to the role of allergy in asthma management as patients in the African American population have been shown to be at greater risk for allergic asthma.

Data will be collected at baseline, 12, and 24 months by telephone interview and from medical records. The hypotheses of the research are that women in the intervention group when compared to the control group will:

* Use emergency department services for asthma less frequently and need urgent care in a physician's office less often;
* Be hospitalized for asthma less frequently.
* Experience fewer symptoms of asthma;
* Have higher levels of asthma-related quality of life

The intervention aims to reduce the burden of asthma as carried by a large subgroup of the adult population. It employs state of the art asthma management strategies and creative means to reach and help patients at high risk of asthma exacerbations and health care use.

ELIGIBILITY:
Inclusion Criteria:

The study participants will be a non-institutionalized ambulatory sample of women who are willing to participate in the project and meet the following criteria:

* Self-identify as African-American
* 18 years of age or older
* Are listed on the University of Michigan Health System (UMHS) Asthma Patient Registry, a validated, all-payer registry of patients with persistent asthma cared for within the UM Health System
* Have access to a telephone or cell phone
* Are not pregnant.. Because the UMHS Asthma Patient Registry is validated, there is minimal risk of diagnostic misclassification. The Registry is created and maintained with a two-step process of identification and validation. UMHS patients with persistent asthma are initially identified through the electronic medical record using National Committee for Quality Assurance (NCQA) Healthcare Effectiveness Data and Information Set (HEDIS) criteria, billing and claims data (when available), and then are validated using documented clinical diagnoses, pulmonary function test (PFT) results, or clinician review.

Exclusion Criteria:

* Patients with chronic respiratory conditions, including cystic fibrosis and chronic obstructive pulmonary disease (COPD) are excluded

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2010-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Emergency department visits - 1st time point | 12months prior to baseline interview
  We will collect health care utilization data related to asthma. Women in the study will be asked during their baseline telephone interview to provide information regarding the frequency of Emergency Department visits related to asthma during the year prior to the baseline interview. Second, women's CareWeb and billing records will be reviewed for asthma related ED visits during this time period.
Emergency Department Visits -2nd time point | Interval between baseline interview and 12 month interview
  We will collect health care utilization data related to asthma. Women in the study will be asked during the SECOND TELEPHONE INTERVIEW to provide information regarding the frequency of Emergency Department visits related to asthma for their year between their baseline and 12month interview. In addition, we will review their CareWeb and billing record data for that time period to see if there are any asthma related Emergency Department visits.
Emergency Department Visits - 3rd time point | Interval between 12 month and 24 month telephone interview
  We will collect health care utilization data related to asthma. Women in the study will be asked during the THIRD TELEPHONE INTERVIEW to provide information regarding the frequency of Emergency Department visits related to asthma for their year between their 12 month and 24 month telephone interview. In addition, we will review their CareWeb and billing record data for that time period to see if there are any asthma related Emergency Department visits.

SECONDARY OUTCOMES:
Hospitalizations - first time point | Year prior to baseline interview
  Women participating in the study will be asked during their BASELINE telephone interview to provide information on hospitalizations related to asthma for the year prior to their baseline interview.In addition, women's Careweb and billing records will be reviewed for hospitalizations for the above mentioned time period.
Hospitalizations related to asthma - 2nd time point | interval between baseline and 12 month interview
  Women participating in the study will be asked during each of their telephone interviews to provide information on hospitalizations related to asthma. During their SECOND TELEPHONE INTERVIEW they will be asked to provide this information for the year between when their baseline interview was conducted and when we are administering the 12 month interview. In addition, women's Careweb and billing records will be reviewed for hospitalizations for the above mentioned time period.
Hospitalizations related to asthma - 3rd time point | interval between 12month and 24 month telephone interview
  Women participating in the study will be asked during each of their telephone interviews to provide information on hospitalizations related to asthma. During their THIRD TELEPHONE INTERVIEW women will be asked to report the number of hospitalizations related to asthma that occurred for the year between when we conducted their 12 month interview and when we are administering the 24month interview. In addition, women's Careweb and billing records will be reviewed for hospitalizations for the above mentioned time period.

CONTACTS AND LOCATIONS:
Overall Officials: Noreen M. Clark, PhD, Principal Investigator — University of Michigan School of Public Health
Locations (1):
- University of Michigan School of Public Health, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Patel MR, Song PX, Sanders G, Nelson B, Kaltsas E, Thomas LJ, Janevic MR, Hafeez K, Wang W, Wilkin M, Johnson TR, Brown RW. A randomized clinical trial of a culturally responsive intervention for African American women with asthma. Ann Allergy Asthma Immunol. 2017 Feb;118(2):212-219. doi: 10.1016/j.anai.2016.11.016. Epub 2016 Dec 27. PMID 28034579
- [Derived] Janevic MR, Sanders GM, Thomas LJ, Williams DM, Nelson B, Gilchrist E, Johnson TR, Clark NM. Study protocol for Women of Color and Asthma Control: a randomized controlled trial of an asthma-management intervention for African American women. BMC Public Health. 2012 Jan 24;12:76. doi: 10.1186/1471-2458-12-76. PMID 22272780